CLINICAL TRIAL: NCT04109625
Title: Preliminary Validation of the Demonstrator of an In Vitro Diagnostic Device for Hepatitis B Screening
Brief Title: Preliminary Validation of an in Vitro Diagnosis-medical Device for Hepatitis B Screening
Acronym: DiVHeB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: MagIA Diagnostics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 38RC.19.159
Record Dates: First submitted 2019-09-20; First posted 2019-09-30 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Hepatitis B; Healthy; Diagnoses Disease
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Intervention Model Description: 3 parallel groups of 10 volunteers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Non-immunized Hepatitis B (Experimental): subjects non-immunized against hepatitis B (naive)
  Interventions: Diagnostic Test: Demonstrator MAGIA
- Vaccine Hepatitis B (Experimental): subjects vaccinated against hepatitis B
  Interventions: Diagnostic Test: Demonstrator MAGIA
- Ongoing, Old or cured Hepatitis B (Experimental): subjects with hepatitis B (old or cured)
  Interventions: Diagnostic Test: Demonstrator MAGIA

INTERVENTIONS:
Diagnostic Test: Demonstrator MAGIA — test of capillary blood with the demonstrator at two time and 2 measures and 2 finger by subject.
  Other Names: v0.1

SUMMARY:
The principal objective of the study is to perform a first step of technical adjustment and preliminary validation of a diagnostic test for hepatitis B (HBsAntigen, anti-HBs Antibody and anti-HBc Antibody) on capillary blood with the device under study in non-immunized subjects against hepatitis B, in subjects with hepatitis B, in subjects with old or cured hepatitis B and in hepatitis B vaccine recipients, compared with the values obtained with the reference technique of medical biology laboratory on serum. The analysis will be performed on the entire cohort.

DETAILED DESCRIPTION:
The diagnosis of hepatitis B in precarious populations is often difficult. The use of a in vitro diagnosis-medical device in point of care could alleviate this difficulty. It would identify whether or not the subjects are infected with the virus, whether they are immunized or not. Then, depending on the results, the subjects could be directly vaccinated or referred to a laboratory of medical biology for confirmation / invalidation of the diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Group 1: HBsAg negative, Anti HBc negative, Anti HBs negative, during a laboratory assay on serum
* Group 2: HBsAg negative, Anti HBc negative, Anti HBs positive, during a laboratory assay on serum
* Group 3: HBsAg negative, Anti HBc positive, Ab anti HBs positive or negative, during a laboratory assay on serum
* Group 4: HBsAg positive, Anti HBc positive, Anti HBs negative, during a laboratory assay on serum
* all: affiliated to social security or beneficiary of such a scheme

Exclusion Criteria:

* Infection by a confounding factor: HIV, HCV and / or HDV
* Protected person: Pregnant woman, parturient, mother who is breastfeeding, person deprived of liberty by judicial or administrative decision, person subject to a legal protection measure
* Exclusion period for other research studies involving the human person
* Annual threshold of allowances for participation in research involving the affected human person.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2022-05-13 (Actual)

PRIMARY OUTCOMES:
feasibility of correlation | Day 0
  To evaluate the feasibility estimated by correlation of the measurements (HBsAg, anti-HBs Ab, HBc-Ab) between the IVD-MD in point of care on capillary blood study and the laboratory results obtained on serum

SECONDARY OUTCOMES:
repeatability of the measurement HBsAg, anti-HBs Ab, HBc-Ab | day 0
  Comparison of the repeatability of the measurement of HBsAg, anti-HBs Ab, HBc-Ab on 2 different fingers with the same device and the same batch of consumables with 2 different times
reproductibility of the measurement HBsAg, anti-HBs Ab, HBc-Ab | day 0
  Comparison of the reproducibility of HBsAg, anti-HBs Ab, HBc-Ab via a test from 2 drops of blood on 2 different fingers with 2 different cartridges and two different readers
correlation according to status | day 0
  Comparison of the correlation coefficients of the measurements between the IVD-MD in point of care and the biology automaton according to the different statuses

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc CRACOWSKI, MD, PhD, Principal Investigator — Grenoble Alps University Hospital
Locations (1):
- Clinical research center CIC1406, Grenoble, France

IPD SHARING:
Plan to Share IPD: Undecided